CLINICAL TRIAL: NCT05622084
Title: Inperia Advance Carbostent™ for Infra-popliteal Artery Stenosis. Evaluation of Safety and Performance in Everyday Clinical Practice: The Inperia Advance Post-Market Retrospective Study
Brief Title: The Inperia Advance Post-Market Retrospective Study
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: CID S.p.A. (Industry)
Collaborators: Meditrial Europe Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: P32203
Record Dates: First submitted 2022-11-11; First posted 2022-11-18 (Actual); Last update posted 2022-11-18 (Actual); Status verified 2022-11

CONDITIONS: Peripheral Arterial Disease
MeSH Terms: conditions — Peripheral Arterial Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Inperia Advance — Patients with infra-popliteal artery stenosis implanted with at least one Inperia Advance device

SUMMARY:
The Inperia Advance Carbostent™ is a CE-marked infra-popliteal stent for treatment of infra-popliteal artery stenosis. The aim of this post-market retrospective study protocl P32203 is to collect clinical data of patients treated with Inperia Advance for the treatment of infra-popliteal artery stenosis in routine clinical practice. In order to obtain long-term follow-up data, the data collection will be limited to patients that have been treated with the device at least 12 months prior to the study start.

DETAILED DESCRIPTION:
The objective of this post-market study is to systematically collect retrospective clinical data on the implantable medical device Inperia Advance in the daily clinical practice in an unselected population treated within the intended use. Data will be collected via medical chart review in anonymous form to assess the safety and efficacy of Inperia Adavance. The Inperia Advance Carbostent™ is a CE-marked infra-popliteal stent for treatment of infra-popliteal artery stenosis.

ELIGIBILITY:
Inclusion Criteria:

* Patient has been implanted with at least one Inperia Advance device according to the indications described in the Instructions for Use (IFU).
* Study device implantation date is at least one year (12 months) prior to the starting date of the retrospective anonymous data collection.

Exclusion Criteria:

* Patients treated less than 12 months prior to study start

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients implanted with at least one Inperia Advance stent for treatment of infra-popliteal artery stenosis, at least 12 months prior to the start date of the retrospective data collection.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2023-02 (Estimated); Primary Completion 2023-06 (Estimated); Study Completion 2023-07 (Estimated)

PRIMARY OUTCOMES:
Rate of Major Adverse Events (MAE) | 12 months
  Composite endpoint of all causes of death, unplanned target limb major amputation and/or clinically indicated target lesion revascularization (TLR)

SECONDARY OUTCOMES:
Primary patency | 6 months and 12 months
  Primary patency is defined as absence of clinically-driven target lesion revascularization or binary restenosis. Binary restenosis is defined as a peak systolic velocity ratio (PSVR) >2.4 (Duplex Ultrasound evaluation)
Limb-salvage rate (LSR) | 6 months and 12 months
  Limb-salvage rate (LSR) is defined as rate of patients free from major amputation. Major amputation is defined as at or above ankle, as opposed to minor amputation being at or below metatarsus preserving functionality of foot
Secondary patency | 6 months and 12 months or latest patency data available
  Patency following successful target lesion revascularization (TLR)
Death | 30 days
  Death within 30 days of the index procedure
Clinically driven Target Lesion Revascularization | 6 months and 12 months
  Clinically driven Target Lesion Revascularization
Target limb ischemia | 6 months and 12 months
  Target limb ischemia requiring surgical intervention or surgical repair of target vessel rate
Rutherford category measurement | pretreatment, 6 months and 12 months
  Rutherford category measurement
Evaluation of Serious Adverse Events (SAEs) | 6 months and 12 months
  Evaluation of Serious Adverse Events (SAEs)
Acute success (device and procedural) within discharge | 24/72 hours
  Clinical device success defined as successful delivery and deployment of the stent(s) at the intended target lesion (this includes successful delivery and deployment of multiple stents) and final residual stenosis of the target lesion minor or equal to 30%, assessed by visual estimation and clinical device success without the occurrence of MAE during the hospital stay

CONTACTS AND LOCATIONS:
Locations (1):
- CHRU Strasbourg, Strasbourg, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Manufactured website — http://www.alvimedica.com/
- See also: Clinical Research Organization — http://www.meditrial.net/